CLINICAL TRIAL: NCT06781931
Title: DG1 Spectacle Lens for Myopia Progression Control in Children: A Three-year Multicenter, Prospective, Randomized, Double-masked, Controlled Clinical Trial to Evaluate the Efficacy and Safety Followed by a One-year Rebound Evaluation
Brief Title: DG1 Spectacle Lens for Myopia Progression Control in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HOYA Lens Thailand LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DG1-101-KIND
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- DG1 Spectacle Lens (Experimental)
  Interventions: Device: DG1 Spectacle Lens
- Single Vision Spectacle Lens (Sham Comparator)
  Interventions: Device: Single Vision Spectacle Lens

INTERVENTIONS:
Device: DG1 Spectacle Lens — DG1 spectacle lens, daily wear for 36 months
  Arms: DG1 Spectacle Lens
Device: Single Vision Spectacle Lens — Single vision spectacle lens, daily wear for 36 months
  Arms: Single Vision Spectacle Lens

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of the DG1 spectacle lens for myopia progression control in children.

* To assess if the DG1 lens will slow the progression of myopia through an adjusted mean difference (e.g., age and baseline SER) of approximately 0.75D in cycloplegic spherical equivalent autorefraction refractive error compared to single-vision (SV) spectacles over the study period.
* To assess if DG1 lens will slow the progression of myopia through an adjusted mean difference (e.g., age and baseline SER) of approximately 0.3mm in axial elongation compared to SV over the study period.

The clinical trial will compare DG1 spectacle lens to single vision spectacle lens.

Participants will wear spectacle lenses and return for visits at regularly scheduled intervals through a 36-month follow up visit. All subjects who complete the 36-month visit will continue in the study for an additional 12 months for the rebound evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject and parent (or guardian) able and willing to provide assent and consent respectively.
2. The subject and parent (or guardian) must attend required study visits and adhere to study requirements.
3. Parent (or guardian) understands and accepts random allocation of grouping, and that subject and parent (or guardian) will not be told the group which the subject is randomized to.
4. The subject is able and willing to wear provided frames and lenses (spectacles), for an average of 10 hours per day for the entirety of the study.
5. Age of subject at time of parent (or guardian) consent and subject assent: 7 to 10 years old (inclusive).
6. Cycloplegic autorefraction spherical equivalent refraction (SER): -1.00 to -5.00 D in each eye at the screening visit.
7. Cycloplegic autorefraction astigmatism of 1.50 D or less in each eye at the screening visit.
8. Cycloplegic spherical equivalent autorefraction (SER) anisometropia of 1.50 D or less at the screening visit.
9. Monocular cycloplegic best corrected distance visual acuity (BCDVA) equal to or better than log MAR 0.10 in each eye at the screening visit.

Exclusion Criteria:

1. Subjects with allergy to fluorescein, benoxinate, proparacaine, cyclopentolate or tropicamide eye drops.
2. Subjects with ocular or systemic abnormalities that might be expected to affect visual functions or refractive development.
3. Subjects who have received treatment of myopia control pharmaceutical medication (e.g., atropine), myopia control contact lenses, other myopia control spectacles, orthokeratology lenses, progressive addition lenses, bifocal lenses, or single vision contact lens prior to entry into the study or during the duration of the study.
4. Subjects with, or a medical history of, strabismus.
5. Subjects with a medical history of binocular vision abnormalities or accommodation abnormalities based on the opinion of the investigator.
6. Subjects with, or history of, amblyopia.
7. Subjects who have participated in a clinical trial within 30 days prior to entry into this study or during participation.
8. Subjects with a history of intraocular surgery.
9. Subjects who, in the judgment of the investigator, have any emotional, physiologic, or anatomical condition which may preclude participation in this study or provide an inappropriate landscape for the intended study treatment.
10. Subjects with pathological myopia (myopia that leads to structural changes in the posterior segment of the eye including posterior staphyloma, myopic maculopathy, and high myopia-associated optic neuropathy).
11. Individuals from the same household (i.e., siblings), employees (or family members of employees) of the Principal Investigator/site, employees (or family members of employees) of the Sponsor, and non-readers.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Co-Primary Effectiveness Endpoints: Spherical equivalent refraction and Axial Length | 36 months
  * The mean difference of cycloplegic autorefractive error progression of the test device as compared to control SV spectacles.
  * The mean difference in axial elongation of the test device as compared to control SV spectacles.

SECONDARY OUTCOMES:
Corrected Visual Acuity | 24 months
  To assess if the DG1 lens will provide a Corrected Visual Acuity (both distance and near) that is no worse than the SV lens with a non-inferiority margin of 10 letters, or 0.2 LogMar (at screening, 12-months and 24-months, compared to their corresponding lens delivery visit).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Irvine Vision Center, Irvine, California
  - Columbia Eye Associates & Family Focus Eye Care, Gainesville, Florida
  - Coan Eye Care and Optical Boutique, Ocoee, Florida
  - Illinois College of Optometry, Chicago, Illinois
  - Complete Eye Care of Medina, Medina, Minnesota
  - Oculus Research, Inc., Garner, North Carolina
  - ProCare Vision Centers, Inc., Granville, Ohio
  - EyeCare Professionals of Powell, Powell, Ohio
  - Southern College of Optometry, Memphis, Tennessee
  - Virginia Pediatric Eye Center, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No